CLINICAL TRIAL: NCT05273931
Title: Evaluation of a Lifestyle Intervention Among Participants of the French Colorectal Cancer Screening Program (LIFE-SCREEN Pilot)
Brief Title: Lifestyle Intervention After Colonoscopy (LIFE-SCREEN Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LIFE-SCREEN pilot
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Higher risk; Lifestyle intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention (Experimental): Lifestyle intervention among participants of the French colorectal cancer screening program
  Interventions: Other: Lifestyle intervention

INTERVENTIONS:
Other: Lifestyle intervention — Documents explaining the strategies to achieve and maintain recommended behaviours as part of a healthier lifestyle

SUMMARY:
The study aims to evaluate the impact of promoting advice on the latest evidence-based diet and lifestyle recommendations for cancer prevention at colorectal cancer (CRC) screening among individuals who may be at higher risk for developing CRC. The overall aim of this LIFE-SCREEN pilot study is to test the trial methods and procedures to be used in the LIFE-SCREEN cluster randomized RCT, in order to discover obstacles and problems prior to the main RCT so that corrective actions can be taken to improve the research process.

The patients (n=40) will be recruited at the Centre Léon Bérard and at the Hôpital Edouard Herriot at the time of CRC screening.

After inclusion, the intervention material (documents explaining the strategies to achieve and maintain recommended behaviours as part of a healthier lifestyle) may be given to the patient during the pre-colonoscopy consultation and/or at the post-colonoscopy visit. Weight, height and blood pressure will be measured during the pre-colonoscopy consultation. Patients will be invited to complete a baseline questionnaire to collect information on their lifestyle, state of health and socio-demographic status. Approximately four to six weeks after, patients will also be asked to complete an evaluation questionnaire asking for their opinion on this material and the procedures. Focus groups with available and willing participants and hospital staff will be organized at the end of the pilot phase recruitment, to gather additional information on the intervention procedures. In addition, all hospital staff will be asked to complete an assessment questionnaire.

Biological samples will then also be collected to test the objective baseline measure of nutritional changes used in the RCT. In order to assess the feasibility and the acceptability of urine, faecal and blood sample collection in this population, the first ten participants recruited (n=10) will be given the option to refuse one or more of the biological sample collections (phase I). Participants will also be asked to complete a questionnaire to provide information on their opinion and willingness to donate biological samples. This assessment questionnaire will allow us to refine the strategies for the other 30 participants (phase II). In this phase II, biological samples will be compulsory (phase IIa) or optional (phase IIb) for all 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* 35-74 years of age
* At increased risk for developing colorectal cancer (CRC), defined here as having a positive faecal immunochemical test (FIT), or family history or symptoms for CRC and identified adenomas but CRC negative during the colonoscopy
* Volunteer and available to get involved in the project throughout the duration of the study,
* Be able to provide informed consent
* Having health insurance (Affiliated to the French social security)
* Score on the adherence to the WCRF recommendations lower or equal to 6 out of 9 (the WCRF score will be assessed based on a short lifestyle questionnaire, annex 1)
* Able to read, write and understand French language

Exclusion Criteria:

* On a strict diet such as meal replacements, diets for co-morbidities such as diabetes
* Lacking mobility due to physical constraints (e.g. handicap that is not compatible with physical activities, uncontrolled cardiovascular diseases/hypertension)
* Planned extensive intestinal surgery such as colectomy or surgical resection of the colon
* Chronic gastrointestinal illness (IBD, IBS, celiac disease)
* Use of any systemic antibiotics, antifungals, antivirals, or antiparasitics in the past 3 months
* Use of probiotic medications in the past 3 months
* History or existence of a primary cancer (apart from an in-situ cancer whatever the location and / or of a cutaneous basal cell cancer and / or of a CRC in complete remission for more than 5 years)
* In a state of severe malnutrition, either:

  ≥10% weight loss in 1 month or ≥ 15% in 6 months
* Cannot be followed for medical, social, family, geographic or psychological reasons, throughout the duration of the study
* Deprived of liberty by court or administrative decision
* Pregnant (for women)
* Concomitant participation in another study on lifestyle
* Optimal lifestyle habits (WCRF score >6) will also be excluded from the pilot study as this participants are not part of target population that could benefit significantly from lifestyle advice (short screener will be completed by patients while in waiting room for pre-colonoscopy visit).

Patients who will be positive for CRC (histological confirmation after colonoscopy) will end prematurely the study.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in adherence to the lifestyle recommendations between baseline and the 4 week follow-up | Change between Baseline and Week 4
  Adherence to the lifestyle recommendations will be measured by the WCRF questionnaire (Diet and Physical Activity)

CONTACTS AND LOCATIONS:
Overall Officials: Anne CATTEY-JAVOUHEY, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Hôpital Edouard Herriot (HCL), Lyon

IPD SHARING:
Plan to Share IPD: No